CLINICAL TRIAL: NCT04678271
Title: Assessment, Feedback, Incentive, Exchange (AFIX-OB) A Customizable Quality Improvement Intervention to Increase Maternal Vaccine Uptake
Brief Title: Assessment, Feedback, Incentive, Exchange (AFIX OB) A Customizable Quality Improvement Intervention to Increase Maternal Vaccine Uptake
Acronym: AFIX-OB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000027357; 1U01IP001110-01 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Influenza; Whooping Cough
Keywords: Pregnancy; Vaccination; Vaccine Acceptance; Influenza; Pertussis; Tdap
MeSH Terms: conditions — Influenza, Human; Whooping Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AFIX-OB Intervention Arm (Experimental): Practices randomized to this arm will choose from a suite of quality improvement interventions that address patient, provider, and practice-level factors relating to maternal vaccination.
  Interventions: Behavioral: AFIX-OB Quality Improvement Package
- Control Arm (No Intervention): Practices randomized to this arm will continue to provide their normal standard of care to pregnant patients at their practice.

INTERVENTIONS:
Behavioral: AFIX-OB Quality Improvement Package — Practices randomized to the intervention arm will be provided with a package of core and supplemental quality improvement interventions to choose from so that the most effective combination for their practice is implemented. Each practice will be required to implement a tablet-based educational app for patients, and evidence based online educational module for providers, standing order protocol, and a reminder/recall protocol. They can then choose to also use flyers and posters in their waiting rooms, standardized talking points for maternal immunization for the providers, educational content for the practice website, and laminated and highlighted CDC Vaccine Information Sheets. The recruited patients and providers at the practice will be given a baseline and follow-up survey to assess their knowledge, attitudes, and beliefs towards maternal immunization.
  Arms: AFIX-OB Intervention Arm

SUMMARY:
The purpose of this study is to evaluate the AFIX-OB model to determine its impact on the change in flu and pertussis (Tdap) uptake, provider knowledge, attitudes and beliefs, and patient knowledge, attitudes and beliefs regarding maternal vaccination. The structure of the model and quality improvement interventions are guided by theory including the elaboration likelihood model and P3 model. These quality improvement measures will be implemented in OB clinics within the Yale New Haven Health System.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-50 years of age
* Currently pregnant and gestational age <26 weeks

Exclusion Criteria:

* Already enrolled in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Influenza Uptake | Baseline and one year after implementation
  Immunization rates for each practice will be collected through JDAT or a random chart review.
Change in Maternal Tdap Uptake | Baseline and one year after implementation
  Immunization rates for each practice will be collected through JDAT or a random chart review.

SECONDARY OUTCOMES:
Change in Patient Vaccine Knowledge | Baseline and one year after implementation
  Data on patient knowledge regarding vaccines will be collected from enrolled participants at the beginning of the study and following the implementation of the intervention via a 10-15 minute survey.
Change in Provider Vaccine Knowledge | Baseline and one year after implementation
  Providers in both study arms will complete baseline and follow-up surveys pre-and post-intervention.
Change in Patient Vaccine Attitudes | Baseline and one year after implementation
  Data on patient attitudes regarding vaccines will be collected from enrolled participants at the beginning of the study and following the implementation of the intervention via a 10-15 minute survey.
Change in Patient Vaccine Beliefs | Baseline and one year after implementation
  Data on patient beliefs regarding vaccines will be collected from enrolled participants at the beginning of the study and following the implementation of the intervention via a 10-15 minute survey.
Change in Provider Vaccine Beliefs | Baseline and one year after implementation
  Providers in both study arms will complete baseline and follow-up surveys pre-and post-intervention.
Change in Provider Vaccine Attitudes | Baseline and one year after implementation
  Providers in both study arms will complete baseline and follow-up surveys pre-and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LeBaron CW, Mercer JT, Massoudi MS, Dini E, Stevenson J, Fischer WM, Loy H, Quick LS, Warming JC, Tormey P, DesVignes-Kendrick M. Changes in clinic vaccination coverage after institution of measurement and feedback in 4 states and 2 cities. Arch Pediatr Adolesc Med. 1999 Aug;153(8):879-86. doi: 10.1001/archpedi.153.8.879. PMID 10437765
- [Background] Chamberlain AT, Seib K, Ault KA, Rosenberg ES, Frew PM, Cortes M, Whitney EA, Berkelman RL, Orenstein WA, Omer SB. Improving influenza and Tdap vaccination during pregnancy: A cluster-randomized trial of a multi-component antenatal vaccine promotion package in late influenza season. Vaccine. 2015 Jul 9;33(30):3571-9. doi: 10.1016/j.vaccine.2015.05.048. Epub 2015 Jun 1. PMID 26044495
- [Background] Dini EF, Chaney M, Moolenaar RL, LeBaron CW. Information as intervention: how Georgia used vaccination coverage data to double public sector vaccination coverage in seven years. J Public Health Manag Pract. 1996 Winter;2(1):45-9. doi: 10.1097/00124784-199600210-00008. PMID 10186655
- [Background] Fairbrother G, Hanson KL, Friedman S, Butts GC. The impact of physician bonuses, enhanced fees, and feedback on childhood immunization coverage rates. Am J Public Health. 1999 Feb;89(2):171-5. doi: 10.2105/ajph.89.2.171. PMID 9949744
- [Background] Frew PM, Murden R, Mehta CC, Chamberlain AT, Hinman AR, Nowak G, Mendel J, Aikin A, Randall LA, Hargreaves AL, Omer SB, Orenstein WA, Bednarczyk RA. Development of a US trust measure to assess and monitor parental confidence in the vaccine system. Vaccine. 2019 Jan 7;37(2):325-332. doi: 10.1016/j.vaccine.2018.09.043. Epub 2018 Nov 30. PMID 30503657
- [Background] Kahn KE, Black CL, Ding H, Williams WW, Lu PJ, Fiebelkorn AP, Havers F, D'Angelo DV, Ball S, Fink RV, Devlin R. Influenza and Tdap Vaccination Coverage Among Pregnant Women - United States, April 2018. MMWR Morb Mortal Wkly Rep. 2018 Sep 28;67(38):1055-1059. doi: 10.15585/mmwr.mm6738a3. PMID 30260946
- [Background] Yuen CY, Tarrant M. Determinants of uptake of influenza vaccination among pregnant women - a systematic review. Vaccine. 2014 Aug 6;32(36):4602-13. doi: 10.1016/j.vaccine.2014.06.067. Epub 2014 Jul 2. PMID 24996123
- [Background] Myers KL. Predictors of maternal vaccination in the United States: An integrative review of the literature. Vaccine. 2016 Jul 25;34(34):3942-9. doi: 10.1016/j.vaccine.2016.06.042. Epub 2016 Jun 18. PMID 27317458
- [Background] Ellingson MK, Dudley MZ, Limaye RJ, Salmon DA, O'Leary ST, Omer SB. Enhancing uptake of influenza maternal vaccine. Expert Rev Vaccines. 2019 Feb;18(2):191-204. doi: 10.1080/14760584.2019.1562907. Epub 2019 Jan 28. PMID 30587042
- [Background] O'Leary ST, Pyrzanowski J, Brewer SE, Dickinson LM, Dempsey AF. Evidence-based vaccination strategies in obstetrics and gynecology settings: Current practices and methods for assessment. Hum Vaccin Immunother. 2016 Apr 2;12(4):866-71. doi: 10.1080/21645515.2015.1130194. PMID 26829978

DOCUMENTS (1):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT04678271/Prot_000.pdf